CLINICAL TRIAL: NCT03380442
Title: Psilocybin and Depression - Assessing the Long-term Effects of a Single Administration of Psilocybin on the Psychiatric Symptoms and Brain Activity of Patients With Severe Depression
Brief Title: Psilocybin and Depression
Acronym: Psilo101
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Helsinki (Other)
Collaborators: Dr. Tomi Rantamäki, Laboratory of Neurotherapeutics, Department of Biosciences, University of Helsinki (Unknown); Dr. Robin Carthart-Harris and Prof. David Nutt, Imperial College London, UK (Unknown)
Responsible Party: Principal Investigator, Jesper Ekelund, Professor of Psychiatry, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2016-004195-22
Record Dates: First submitted 2017-12-12; First posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Severe Depression
Keywords: fMRI; psilocybin; ketamine; biomarker; rapid-acting antidepressants
MeSH Terms: conditions — Depression | interventions — Psilocybin; Ketamine

STUDY DESIGN:
Intervention Model Description: In a randomized, double-blind placebo-controlled design, 20 of the participants will receive ketamine, and 20 will receive psilocybin. 20 of the participants will be included in the study as a no-treatment group, so that natural time-dependent changes in depressive symptoms can be controlled for and thus the antidepressive effects of ketamine and psilocybin treatment can be verified. The no-treatment group will only attend the initial clinical interviews, and their depressive symptoms will be assessed remotely.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Since the psilocybin is ingested orally in capsule form, whereas ketamine is administered intranasally, the participants will either receive a placebo capsule containing microcrystalline cellulose (if they belong to the group receiving ketamine), or intranasally administered saline solution (with added bitter flavoring which will mimic the taste of ketamine that is often detectable even when administered intranasally).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Psilocybin group (Experimental): This group will receive a single oral 25mg dose of psilocybin under surveilled and safe conditions.
  Interventions: Drug: Psilocybin
- Ketamine group (Active Comparator): This group will receive a single intranasal 125mg dose of ketamine under surveilled and safe conditions.
  Interventions: Drug: Ketamine (Ketalar)
- No-treatment group (No Intervention): This group will be included in the study as a no-treatment group, so that natural time-dependent changes in depressive symptoms can be controlled for and thus the antidepressive effects of ketamine and psilocybin treatment can be verified

INTERVENTIONS:
Drug: Psilocybin — Psilocybin ingested orally
  Arms: Psilocybin group
Drug: Ketamine (Ketalar) — Ketamine administered intranasally
  Arms: Ketamine group

SUMMARY:
The main aim of the study is to investigate the possible long-term therapeutic effects of psilocybin on the symptoms of severe depression, as well as the brain mechanisms underlying these changes. Depression severity is assessed before and after (i.e., 1 week, 3 months and 6 months after) a single dose of psilocybin and compared to respective scores of a group receiving an active placebo, ketamine. Brain activity (using functional magnetic resonance imaging) is measured before and one week after drug administration in order to determine whether changes in brain networks related to emotional and self-referential processing correlate with any observed changes in depression scores. Further, blood samples will be obtained from the participants and analyzed in order to reveal gene expression and molecular level correlates underlying rapid antidepressant effects, and to identify biomarkers that predict treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Major depression of a moderate to severe degree (17+ on the 21-item HAM-D).
2. No health-related contraindications.

Exclusion Criteria:

1. Current or previously diagnosed psychotic disorder.
2. Immediate family member with a diagnosed psychotic disorder.
3. Medically significant condition rendering unsuitability for the study (e.g., diabetes, epilepsy, severe cardiovascular disease, hepatic or renal failure etc.).
4. History of suicide attempts.
5. History of mania.
6. Current 5-HT2A antagonist antidepressant medication.
7. Blood or needle phobia.
8. Positive pregnancy test.
9. Current drug or alcohol dependence.
10. Lack of appropriate use of contraception.
11. Breast-feeding.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
The 16-Item Quick Inventory of Depressive Symptomatology (QIDS) | 6 months
  The primary outcome measures in this study will be the mean change in QIDS scores from pre-administration baseline at day 1 to Follow-up 2 at day 103 (3 months after the administration session). Additionally, an electronic version of the QIDS will be performed 6 months after the administration session. The criteria for determining response will be a reduction of 25% in the (QIDS; Rush et al., 2003) scores from baseline (screening), and remission will be scores of ≤5 on the QIDS.

SECONDARY OUTCOMES:
The Montgomery and Asberg Depression Rating Scale | 3 months
  The Montgomery and Asberg Depression Rating Scale will be carried out at screening ( day 1), Follow-up 1 (day 18) and Follow-up 2 (day 103, 3 months after the administration session).
Hamilton Depression Rating Scale | 3 months
  The Hamilton Depression Rating Scale will be carried out at screening ( day 1), Follow-up 1 (day 18) and Follow-up 2 (day 103, 3 months after the administration session).

IPD SHARING:
Plan to Share IPD: No